CLINICAL TRIAL: NCT04927078
Title: Analysis of Vital Signs in Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Oxehealth Limited (Industry)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 287454
Record Dates: First submitted 2021-04-13; First posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Respiratory Disease
Keywords: Breathing rate; Pulse rate; COVID 19; Patient monitoring
MeSH Terms: conditions — Respiration Disorders; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with COVID 19 diagnosis: We will measure the breathing rate (BR) before and after the clinical diagnosis of COVID 19.
  Interventions: Other: Observation of breathing pattern
- Participants without COVID 19 diagnosis: Breathing rates will be measured for the same time duration as the cases.
  Interventions: Other: Observation of breathing pattern

INTERVENTIONS:
Other: Observation of breathing pattern — Observations will be collected using a remote vision based patient monitoring and management system.

SUMMARY:
This project will use data obtained from a proprietary vision-based patient monitoring and management system (OxeVision) for measuring heart rate and respiratory rate which is in clinical use at the Coventry and Warwickshire Partnership NHS Trust.

DETAILED DESCRIPTION:
The investigators will analyse data from patients with known COVID 19 infection both during, and where possible before clinical COVID 19 infection and controls to determine whether changes can be detected in these parameters that precede overt clinical deterioration. The role of remote vision-based patient monitoring and management in supporting the care of patients with COVID-19 will be assessed through staff interviews.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 and above. Patients on wards with a medical diagnosis of COVID 19 who are in rooms with the Vision based patient monitoring and management system.

Exclusion Criteria:

Children will be excluded. No data will be excluded unless specifically requested by the treating clinician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants admitted to inpatient mental health wards.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Breathing rates | Data will be collected throughout study completion, an average of 7 months, to obtain breathing rate before and after the diagnosis of COVID 19.
  Breathing rates collected via remote monitoring of participants using the Vision Based Patient Monitoring and Management System.

SECONDARY OUTCOMES:
Pulse rates | Data will be collected throughout study completion, an average of 7 months, to obtain pulse rate before and after the diagnosis of COVID 19.
  Pulse rate collected via remote monitoring of participants using the Vision Based Patient Monitoring and Management System.
BR and PR | Data will be collected throughout study completion, an average of 7 months, to obtain breathing and pulse rate before and after the diagnosis of COVID 19.
  Similar data to be collected from control subjects

CONTACTS AND LOCATIONS:
Overall Officials: Michael Polkey, Principal Investigator — The Royal Bromptom Hospital
Locations (1):
- Coventry and Warwickshire Partnership NHS, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided